CLINICAL TRIAL: NCT05953454
Title: Effectiveness of Group Versus Individual Pain Neuroscience Education on Clinical and Psychosocial Outcomes in Patients With Chronic Low Back Pain: Protocol of a Randomized Controlled Trial
Brief Title: Effectiveness of Pain Neuroscience Education on Clinical and Psychosocial Variables in Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Santo Tomas, Chile (Other)
Responsible Party: Principal Investigator, Joaquín Ignacio Salazar Méndez, adjunct teacher, Universidad Santo Tomas, Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USantoTomasChile
Record Dates: First submitted 2023-07-01; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Chronic Low-back Pain
Keywords: pain neuroscience education; physical therapy; chronic pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Pain Neuroscience Education (Experimental): A single face-to-face group session of approximately 60-80 minutes provided through active participation. Five key domains will be structured from the Fear and Belief Avoidance Questionnaire that will serve as a guide for the sessions through a Powerpoint presentation. In addition, participants will be encouraged to be active by walking for 20-30 minutes 3-5 times a week and will be taught an exercise to improve transverse abdominis activation (abdominal corset or follow-through).
  With the main ones, a brochure will be delivered and informative capsules will be made to which the participants will have access (5 videos of 15 minutes, one per domain). Participants will be instructed to record on a calendar the days they read the brochure and/or reviewed the information capsules to assess treatment compliance and for each domain invent a metaphor or script for how they would explain it to another person. This activity must be delivered in the second evaluation.
  Interventions: Other: Pain neuroscience Education
- Individual Pain Neuroscience Education (Experimental): A single one-on-one face-to-face session of approximately 60-80 minutes provided through active participation. Five key domains will be structured from the Fear and Belief Avoidance Questionnaire that will serve as a guide for the sessions through a Powerpoint presentation. In addition, participants will be encouraged to be active by walking for 20-30 minutes 3-5 times a week and will be taught an exercise to improve transverse abdominis activation (abdominal corset or follow-through).
  With the main ones, a brochure will be delivered and informative capsules will be made to which the participants will have access (5 videos of 15 minutes, one per domain). Participants will be instructed to record on a calendar the days they read the brochure and/or reviewed the information capsules to assess treatment compliance and for each domain invent a metaphor or script for how they would explain it to another person. This activity must be delivered in the second evaluation.
  Interventions: Other: Pain neuroscience Education
- Control (No Intervention): no intervention

INTERVENTIONS:
Other: Pain neuroscience Education — A pain neuroscience education session geared towards fear-avoidance beliefs
  Arms: Group Pain Neuroscience Education; Individual Pain Neuroscience Education

SUMMARY:
An educational intervention on the neurophysiology of chronic pain will be provided. The content of the intervention will be identical in the experimental groups (group and individual). The intervention has an active educational approach based on reconceptualizing the maladaptive beliefs that influence the fear-avoidance behavior of the participants through updated contents of the neuroscience of pain.

The effects of the intervention will be compared between the groups and the influence of the social determinants of health on the effects will also be determined.

The investigators hypothesize that there will be significant differences in favor of the group intervention group over the individual intervention groups. Furthermore, the effects will be influenced by the social determinants of health in both experimental groups.

ELIGIBILITY:
Inclusion Criteria:

* non-specific low back pain ≥ 3 months without compromise of any lower limb.
* average pain intensity ≥ 3/10 and ≤8/10 (according to the 0-10 numerical rating scale [NRS]) in the last month.

Exclusion Criteria:

* psychiatric, neurological or oncological diseases.
* operated of some lumbar pathology
* chronic low back pain due to a specific cause (lumbar stenosis, herniated disc, spinal deformity, fracture, spondylosis)
* have received any modality of active or passive physical therapy for pain in the last two months,
* previous experiences with PNE

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Fear avoidance beliefs | baseline, 1-week post-intervention, and 4 -weeks post-intervention
  The Fear Avoidance Beliefs Questionnaire consists of two subscales: (1) a 7-item work subscale (FABQ-W) and (2) a 4-item physical activity subscale (FABQ-P). Both subscales score on a Likert-type scale from 0 to 6 points on each item. Higher scores indicate higher levels of fear-avoidance beliefs.
changes in pressure pain sensitivity | baseline, 1-week post-intervention, and 4 -weeks post-intervention
  An algometer will be used to measure pressure pain sensitivity (SPD), which is defined as the amount of applied pressure required for a subject to report the onset of pain sensation. It will be applied three times for each moment of evaluation and the average of the three applications will be considered. The unit of measure kg/cm2/s will be used.

SECONDARY OUTCOMES:
Changes in Pain Self-efficacy | baseline, 1-week post-intervention, and 4 -weeks post-intervention
  Cain self-efficacy questionnaire (PSEQ) consists of 10 items rated on a 7-point Likert scale from 0 ("not at all sure") to 6 ("very sure"). Higher scores indicate stronger self-efficacy beliefs, while low scores indicate a subject more focused on their pain.
Changes in Catastrophizing | baseline, 1-week post-intervention, and 4 -weeks post-intervention
  Pain Catastrophizing Scale (PCS) consists of 13 items on a 5-point Likert scale ranging from (0) never to (4) all the time. Higher scores indicate more catastrophic thoughts.
Changes in Pain intensity | baseline, 1-week post-intervention, and 4 -weeks post-intervention
  Numerical Rating Scale (NRS). It consists of a number line from 0 to 10. Higher scores indicate greater intensity of pain.
Treatment expectation | baseline
  The treatment expectation questionnaire (TEX-Q). This questionnaire consists of 15 questions with a Likert scale of 0-10. higher scores indicate a better expectation of treatment.

OTHER OUTCOMES:
Employment status | baseline
  employed versus unemployed
Educational level | baseline
  participants were assigned to the lower educational level if they had not completed secondary education and to the higher educational level if they had completed secondary education or university studies
economic income | baseline
  individual monthly taxable income

CONTACTS AND LOCATIONS:
Overall Officials: Joaquín I Salazar, MSc, Principal Investigator — Universidad Santo Tomás

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: from 6 months after publication. They will be available for one year.
Access Criteria: will be provided to any researcher who requires it via email